CLINICAL TRIAL: NCT04636190
Title: A Retrospectively Enrolled and Prospectively Followed, Post-market, Multi-center Evaluation of the Clinical Outcomes of the Triathlon All-Polyethylene Tibia
Brief Title: Triathlon All-Polyethylene Tibia Outcomes Study
Acronym: APT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-03

CONDITIONS: Arthropathy of Knee; Replacement; Knee Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Triathlon All-Polyethylene Tibia Knee (Other): All subjects enrolled will have received the Triathlon All-Polyethylene Tibia Knee device.
  Interventions: Device: Triathlon All-Polyethylene Tibia Knee

INTERVENTIONS:
Device: Triathlon All-Polyethylene Tibia Knee — Triathlon All-Polyethylene Tibia Knee is an all polyethylene resurfacing knee device using either a condylar stabilizing (CS) and posterior stabilizing (PS) device.

SUMMARY:
The purpose of this study is to evaluate the clinical functional results of the Triathlon All-Polyethylene Tibia Knee Device.

DETAILED DESCRIPTION:
This study is a retrospectively enrolled, prospective evaluation of the Triathlon All-Polyethylene Tibia (APT) for patients who meet the eligibility criteria. The enrolled cases will be followed for outcomes measured to 10 years. A modular, Triathlon metal-backed tibia (MBT) and polyethylene insert construct will be used as a historical control.

ELIGIBILITY:
Inclusions:

* Patient underwent primary TKA and is currently implanted with the Triathlon All- Polyethylene Tibia as well as compatible Stryker femoral and patellar components with no pending revision or removal.
* Patient has signed an IRB-approved, study specific Informed Patient Consent Form.
* Patient is a male or non-pregnant female and is 18 years of age or older at the time of study device implantation.
* Patient is willing and able to comply with postoperative scheduled clinical and radiographic evaluations.

Exclusions:

* Patient had an active or suspected latent infection in or about the affected knee joint at time of study device implantation.
* Patient had distant foci of infection which could have caused hematogenous spread to the implant site at time of study device implantation.
* Patient was skeletally immature at time of study device implantation.
* Patient has a mental or neuromuscular disorder which would create an unacceptable risk of prosthesis instability, prosthesis fixation failure, or complications in postoperative care.
* Patient's bone stock was compromised by disease, infection, or prior implantation which cannot provide adequate support and/or fixation to the prosthesis.
* Patient had severe instability of the knee joint secondary to the absence of collateral ligament integrity and function.
* Patient was immunologically suppressed or receiving steroids in excess of normal physiological requirements at the time of surgery (e.g. > 30 days).
* Patient is a prisoner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2033-10 (Estimated); Study Completion 2033-10 (Estimated)

PRIMARY OUTCOMES:
Knee Society Score (KSS) Function | 10-years postoperative
  The Knee Society Clinical Rating System is comprised of two distinct sub-scores: one for pain, range of motion (ROM) and joint stability, and one for functional parameters. Sub-scores range from a potential minimum score of 0 to a maximum score of 100 points. Although the specific scores are not distinguished as "excellent," "good," "fair," or "poor," a higher value represents a better outcome postoperative.

SECONDARY OUTCOMES:
Kaplan-Meier Survival Analysis | 10-years postoperative
  To present 10-year Kaplan-Meier survival analysis for the Triathlon APT

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Michigan Orthopaedic Center, Lansing, Michigan
  - Kaleida Health, Department of Orthopaedic Surgery, Buffalo General Hospital, Buffalo, New York
  - Syracuse Orthopedic Specialists, PC, Syracuse, New York
  - Duke University Medical Center, Durham, North Carolina
  - Department of Orthopaedic Surgery Cleveland Clinic, Cleveland, Ohio
  - Musculoskeletal Institute, University of Texas Health Austin, Austin, Texas